CLINICAL TRIAL: NCT01366339
Title: A Replicate Design, Double-Blind, Randomized, Placebo-Controlled Tolerance and Pharmacokinetics Study of N-Methylnaltrexone Tablets in Normal, Healthy Volunteers
Brief Title: Tolerance and Pharmacokinetics Study of MNTX Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, MD, Progenics Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MNTX 1201
Record Dates: First submitted 2011-05-27; First posted 2011-06-06 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Normal Healthy Volunteers
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): Oral methylnaltrexone
  Interventions: Drug: Oral methylnaltrexone
- Arm 2 (Experimental): Oral methylnaltrexone
  Interventions: Drug: Oral methylnaltrexone
- Arm 3 (Experimental): Oral methylnaltrexone
  Interventions: Drug: Oral methylnaltrexone
- Arm 4 (Placebo Comparator): Oral placebo
  Interventions: Drug: Oral placebo

INTERVENTIONS:
Drug: Oral methylnaltrexone
  Arms: Arm 1; Arm 2; Arm 3
Drug: Oral placebo
  Arms: Arm 4

SUMMARY:
This is a double-blind, randomized, placebo-controlled, phase I study in normal healthy volunteers. Study treatment includes single doses of MNTX and placebo. In addition, half of each active treatment group is further randomized to a second, replicate dose of MNTX, and the placebo group receives an additional placebo dose.

ELIGIBILITY:
Inclusion Criteria:

1. Weight between 55 and 85 kg
2. In good health with no evidence of a clinically significant chronic medical condition
3. Non-Smokers.

Exclusion Criteria:

1. History of asthma, allergic skin rash, significant allergy or other immunologic disorder
2. Known or suspected hypersensitivity to opioids or opioid antagonists
3. History or suspicion of alcohol or drug abuse.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2003-10; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of oral doses of MNTX | 7 days
  To determine PK, dose proportionality, and urinary excretion of single, oral doses of MNTX in normal healthy volunteers

SECONDARY OUTCOMES:
Peak Time of Maximum Concentration (Tmax) of oral doses of MNTX | 7 days
  To determine PK, dose proportionality, and urinary excretion of single, oral doses of MNTX in normal healthy volunteers
Area Under the Plasma Concentration versus Time Curve (AUC) of oral doses of MNTX | 7 days
  To determine PK, dose proportionality, and urinary excretion of single, oral doses of MNTX in normal healthy volunteers
Half-life of oral doses of MNTX | 7 days
  To determine PK, dose proportionality, and urinary excretion of single, oral doses of MNTX in normal healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States